CLINICAL TRIAL: NCT02569905
Title: Tumor Hospital of Guangxi Medical University, China
Brief Title: Effect of Parecoxib Sodium and Flurbiprofen Injection on Postoperative Shivering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, xueke du, anesthesiologists, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014032605
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Shivering
Keywords: flurbiprofen; Parecoxib sodium; Postoperative Shivering
MeSH Terms: interventions — parecoxib; Flurbiprofen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Groups Parecoxib sodium (Active Comparator): Fifty-one, American Society of Anesthesiologists' (ASA) physical status1or2, patients, undergoing colorectal operation were selected in the clinical study.
  Interventions: Drug: parecoxib sodium
- Groups Flurbiprofen (Active Comparator): Fifty-two, American Society of Anesthesiologists' (ASA) physical status1or2, patients, undergoing colorectal operation were selected in the clinical study.
  Interventions: Drug: flurbiprofen
- Group Saline (Placebo Comparator): Fifty-one, American Society of Anesthesiologists' (ASA) physical status1or2, patients, undergoing colorectal operation were selected in the clinical study.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: parecoxib sodium — parecoxib sodium 40mg
  Arms: Groups Parecoxib sodium
Drug: flurbiprofen — flurbiprofen 50mg
  Arms: Groups Flurbiprofen
Drug: saline — normal saline
  Arms: Group Saline

SUMMARY:
Shivering is an early postoperative complication during the postoperative recovery period, and there is no clear consensus about the best way for its prevention. The aim of the study was to compare the efficacy and accompanying side effects of prophylactic flurbiprofen with that of parecoxib or placebo for reducing postoperative shivering.

DETAILED DESCRIPTION:
154 patients with American Society of Anesthesiologists physical status I-II, who were scheduled for colorectal operation under general anesthesia, were randomly assigned to receive flurbiprofen (Group F), parecoxib sodium (Group P ) or normal saline(Group S)40min before the end of surgery. Hemodynamic parameters were monitored. The occurrence of shivering postoperative nausea and vomiting were recorded during the recovery period. And visual analogue score (VAS) and ramsy sedation scale (RSS) were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* One hundred and sixty-six, American Society of Anesthesiologists' (ASA) physical status1or2, patients, undergoing colorectal operation were selected in the prospective, randomized, double-blind clinical study.
* All patients who were from 21 to 62 years old and body mass index 19-35 in tumor hospital of Guangxi medical university (State of China) from April 2014 to April 2015 were included.

Exclusion Criteria:

* Patients with cardiac, pulmonary, hepatic, renal, thyroid, or neuromuscular disease, and those who took chronic drug or abused alcohol were excluded.
* Another patients with hypertension, gastrointestinal bleeding, an initial core temperature >37.5℃ or <36.5℃, a history of allergy to non- steroidal anti-inflammatory drugs (NSAIDs) or other agents to be used, and inability to cooperate were also excluded in this study.
* Another patients with blood loss during operation>400ml, a need for blood transfusion during surgery, duration of operation>4h and surgical procedures changed were excluded.

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
shivering | in one hour after extubation.

SECONDARY OUTCOMES:
visual analogue score | at the time of extubation, 30min and 60min after extubation.
sedation scores | at the time of extubation, 30min and 60min after extubation.
incidence of postoperative nausea and vomiting | in one hour after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Department, Tumor Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Background] Buggy DJ, Crossley AW. Thermoregulation, mild perioperative hypothermia and postanaesthetic shivering. Br J Anaesth. 2000 May;84(5):615-28. doi: 10.1093/bja/84.5.615. No abstract available. PMID 10844839
- [Background] Kilbas Z, Mentes MO, Harlak A, Yigit T, Balkan SM, Cosar A, Ozturk E, Kozak O, Tufan CT. Efficacy of wound infiltration with lornoxicam for postoperative analgesia following thyroidectomy: a prospective, randomized, double-blind study. Turk J Med Sci. 2015;45(3):700-5. doi: 10.3906/sag-1402-125. PMID 26281342
- [Background] Yang X, Peng N, Li N, Li J. Effect of cyclooxygenase-2-specific inhibitors on postoperative analgesia after major open abdominal surgery. Pain Manag Nurs. 2015 Jun;16(3):242-8. doi: 10.1016/j.pmn.2014.07.004. PMID 26025794
- [Background] Ayrian E, Kaye AD, Varner CL, Guerra C, Vadivelu N, Urman RD, Zelman V, Lumb PD, Rosa G, Bilotta F. Effects of Anesthetic Management on Early Postoperative Recovery, Hemodynamics and Pain After Supratentorial Craniotomy. J Clin Med Res. 2015 Oct;7(10):731-41. doi: 10.14740/jocmr2256w. Epub 2015 Aug 23. PMID 26345202
- [Background] Yared JP, Starr NJ, Hoffmann-Hogg L, Bashour CA, Insler SR, O'Connor M, Piedmonte M, Cosgrove DM 3rd. Dexamethasone decreases the incidence of shivering after cardiac surgery: a randomized, double-blind, placebo-controlled study. Anesth Analg. 1998 Oct;87(4):795-9. doi: 10.1097/00000539-199810000-00010. PMID 9768772
- [Background] Li X, Zhou M, Xia Q, Li W, Zhang Y. Effect of parecoxib sodium on postoperative shivering: a randomised, double-blind clinical trial. Eur J Anaesthesiol. 2014 Apr;31(4):225-30. doi: 10.1097/01.EJA.0000436684.94403.1e. PMID 24270900
- [Background] Chen J, Chen Y, Lu KZ. Prophylactic parecoxib reduces the incidence of shivering after general anaesthesia. Eur J Anaesthesiol. 2014 Dec;31(12):714-5. doi: 10.1097/EJA.0000000000000165. No abstract available. PMID 25335108
- [Background] Shen H, Chen Y, Lu KZ, Chen J. Parecoxib for the prevention of shivering after general anesthesia. J Surg Res. 2015 Jul;197(1):139-44. doi: 10.1016/j.jss.2015.03.011. Epub 2015 Mar 28. PMID 25908099
- [Background] Teymourian H, Mohajerani SA, Bagheri P, Seddighi A, Seddighi AS, Razavian I. Effect of Ondansetron on Postoperative Shivering After Craniotomy. World Neurosurg. 2015 Dec;84(6):1923-8. doi: 10.1016/j.wneu.2015.08.034. Epub 2015 Sep 3. PMID 26342782
- [Background] Liu ZX, Xu FY, Liang X, Zhou M, Wu L, Wu JR, Xia JH, Zou Z. Efficacy of dexmedetomidine on postoperative shivering: a meta-analysis of clinical trials. Can J Anaesth. 2015 Jul;62(7):816-29. doi: 10.1007/s12630-015-0368-1. Epub 2015 Apr 8. PMID 25851018
- [Background] Park SM, Mangat HS, Berger K, Rosengart AJ. Efficacy spectrum of antishivering medications: meta-analysis of randomized controlled trials. Crit Care Med. 2012 Nov;40(11):3070-82. doi: 10.1097/CCM.0b013e31825b931e. PMID 22890247